CLINICAL TRIAL: NCT01796145
Title: A Study to Evaluate the Impact of Liver Stiffness on Treatment Outcome of Hepatocellular Carcinoma
Brief Title: Fibroscan Study in HCC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Cancer Trials Unit, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HCC033
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Confirmed Diagnosis of Hepatocellular Carcinoma; Patients Who Are Scheduled to Undergo Transarterial Chemobolization, Systemic Therapy Surgery; Child's A to C Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TACE (Experimental)
  Interventions: Other: Fibroscan
- Systemic Therapy (Experimental)
  Interventions: Other: Fibroscan
- Surgery (Experimental)
  Interventions: Other: Fibroscan

INTERVENTIONS:
Other: Fibroscan

SUMMARY:
In patients with HCC undergoing therapy 1. We aim to determine the prognostic significance of liver stiffness in patients with HCC 2. We aim to determine the rate and severity of complications of treatment and its association with liver stiffness in patients with HCC

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HCC
* Patients who are scheduled to undergo therapy, either TACE systemic therapy or surgery

  1. For TACE cohort, patients undergoing first cycle TACE are eligible.
  2. For systemic therapy cohort, patients undergoing first-line systemic therapy are eligible.
  3. For surgery cohort, patient undergoing surgery are eligible.
* Prior surgery or loco-ablative therapy (e.g. Radiofrequency ablation, microwave, percutaneous ethanol injection) is allowed
* Child's A to Child's C liver function

Exclusion Criteria:

* ECOG performance status > 2
* Poorly controlled ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2013-02-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Rate and grade of treatment complications | 2 years
Liver stiffness (kPa) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam Chan, FHKCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong